CLINICAL TRIAL: NCT01966835
Title: Effect of Moderate to High Intensity Aerobic Interval Training on Polysomnographic Measured Sleep in Patients With Rheumatoid Arthritis. A Randomized Controlled Trial
Brief Title: Effect of Moderate to High Intensity Aerobic Interval Training on Polysomnographic Measured Sleep in Patients With Rheumatoid Arthritis
Acronym: JR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Katrine Loeppenthin, PhD student, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: JR sleep
Record Dates: First submitted 2013-10-16; First posted 2013-10-22 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Rheumatoid Arthritis; Sleep Disturbances
Keywords: sleep quality; sleep disturbances; high intensity aerobic interval training; rheumatoid arthritis; fatigue; pain; polysomnography; watt max
MeSH Terms: conditions — Arthritis, Rheumatoid; Parasomnias; Sleep Initiation and Maintenance Disorders; Fatigue; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High intensity aerobic interval training (Experimental): The intervention consists of a total of 18 moderate-to-high intensity aerobic interval training sessions (20-30 minutes/session) spread over a maximum of eight weeks (2-3 times/week) as shown in Table 1. The training sessions are performed on bicycle ergometers (Kettler) and supervised by physiotherapists. Each session is built up by brief periods of high-intensity aerobic exercise (70-80 %) separated by recovery periods of lower-intensity (40-50%). Each session is introduced by a 5-minute warm-up and ends with a 5-minute cool-down (equivalent to 40-50% watt max). The absolute exercise intensity/workload (watt) is determined individually for each participant based on the watt max test performed at baseline.
  Interventions: Behavioral: High intensity aerobic interval training
- control group (No Intervention): no exercise intervention

INTERVENTIONS:
Behavioral: High intensity aerobic interval training — The intervention consists of a total of 18 moderate-to-high intensity aerobic interval training sessions (20-30 minutes/session) spread over a maximum of eight weeks (2-3 times/week) as shown in Table 1. The training sessions are performed on bicycle ergometers (Kettler) and supervised by physiotherapists. Each session is built up by brief periods of high-intensity aerobic exercise (70-80 %) separated by recovery periods of lower-intensity (40-50%). Each session is introduced by a 5-minute warm-up and ends with a 5-minute cool-down (equivalent to 40-50% watt max). The absolute exercise intensity/workload (watt) is determined individually for each participant based on the watt max test performed at baseline.
  Arms: High intensity aerobic interval training

SUMMARY:
Poor sleep quality and sleep disturbances are common in patients with rheumatoid arthritis and are associated with an increased risk of co-morbidity and all-cause mortality.Few studies have examined the possibilities of improving sleep in patients with rheumatoid arthritis, and the focus has primarily been on medical treatment. Aerobic exercise training constitutes a potentially promising, non-pharmacological alternative to improve sleep.

This study is a randomized controlled trial of 44 patients with rheumatoid arthritis.

The aim is to investigate the effect of a moderate-to-high intensity aerobic interval training intervention on sleep quality and sleep disturbances in patients with rheumatoid arthritis.

The primary hypothesis is that moderate-to high intensity aerobic exercise will improve objective measured sleep quality and sleep disturbances. The secondary hypothesis is that the intervention may improve fitness, subjective sleep quality and physical function as well as reduce pain, fatigue, depressive symptoms and improve health-related quality of life.

DETAILED DESCRIPTION:
Poor sleep quality and sleep disturbances are common in patients with rheumatoid arthritis and are associated with an increased risk of co-morbidity, including cardiovascular diseases, diabetes, hypertension, and all-cause mortality. In addition, poor sleep quality is associated with fatigue, pain and physical disability. Few studies have examined the possibilities of improving sleep in patients with rheumatoid arthritis, and the focus has primarily been on medical treatment. Aerobic exercise training constitutes a potentially promising, non-pharmacological alternative to improve sleep in healthy people and patients with insomnia.

The present study is a blinded randomized controlled trial of 44 patients with a diagnosis of rheumatoid arthritis.

The aim is to examine the effect of an aerobic exercise intervention, consisting of 18 exercise sessions, on sleep quality and sleep disturbances in patients with rheumatoid arthritis who experience poor sleep quality.

The primary hypothesis is that moderate to high intensity aerobic exercise will improve objective measured (by polysomnography) sleep quality and sleep disturbances. The secondary hypothesis is that the intervention may improve fitness, subjective sleep quality and physical function as well as reduce pain, fatigue, depressive symptoms and improve health-related quality of life.

The study will provide evidence on the effect of moderate-to-high-intensity aerobic exercise on the improvement of sleep in patients with rheumatoid arthritis. Specifically, the results are expected to provide important evidence about the potential of interval training to improve quality of sleep and sleep disturbances. As such, the study meets a currently unmet need for non-pharmacological treatment initiatives of poor sleep in patients with a systemic inflammatory disorder.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years
* a clinical diagnosis of rheumatoid arthritis
* Experience poor sleep quality (PSQI >5)
* Low disease activity (DAS28<3.2)
* Understand Danish

Exclusion Criteria:

* Documented sleep apnea (AHI >15/hour)
* ECG that does not allow exercise
* Night work during the period in which the intervention takes place
* Pregnant or are breast-feeding
* Treatment with steroid, hypnotics, antidepressants, antipsychotics
* Cardiac symptoms - NYHA >2
* Regular physically active (aerobic exercise >3 x per week)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
sleep | Change from baseline in objectively measured sleep to 8 weeks
  Measured by polysomnography. Polysomnography is a objective measurement of sleep duration, sleep stages and sleep quality.

SECONDARY OUTCOMES:
Cardiopulmonary fitness | change in baseline in VO2-max to 8 weeks
  The patients' aerobic capacity is assessed by an incremental maximum work test on bicycle ergometer. Following a 5-minute warm-up period on individual steady state work intensity, the work load increases by 20 watt each minute until exhaustion.
Plasma | change from baseline in plasma to 8 weeks
  C-reactive protein (CRP) and hemoglobin are assessed
physiological outcomes | change from baseline in blood pressure, weight and height to 8 weeks
Disease activity | change from baseline in disease activity to 8 weeks
  Disease Activity Score (DAS28) is calculated from the number of swollen and tender joints (28 joints), CRP and the patients' global assessment of arthritis
self reported sleep quality and sleep disturbances | change from baseline in selfreported sleep to 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI) measures self-reported sleep quality and disturbances during the previous four weeks
self reported sleepiness | change from baseline in sleepiness to 8 weeks
  The Epworth Sleepiness Scale measures self-reported daytime sleepiness.
self reported fatigue | change from baseline in fatigue to 8 weeks
  The Bristol Rheumatoid Arthritis Fatigue Multi-Dimensional Questionnaire (BRAF MDQ)measures self-reported fatigue
self reported depressive symptoms | change from baseline in depressive symptoms to 8 weeks
  The Center for Epidemiological Studies-Depression (CES-D) measures self-reported depressive symptoms.
Physical function | change from baseline in HAQ score to 8 weeks
  The Health Assessment Questionnaire (HAQ) measures self-reported physical function.
self reported Health-related quality of life | change from baseline in health related quality of life to 8 weeks
  EuroQol (EQ-5D-5L)measures health-related quality of life.
Health and lifestyle questionnaire | change from baseline in health and lifestyle to 8 weeks
  Information about self-reported comorbidity, age, gender, education, work, income, physical activity, smoking, alcohol and caffeinated drinks per day will be recorded. Patients are also asked of information about actual medical treatment.
Sleep pattern | change from baseline to 8 weeks
  Patients complete sleep diaries for 14 days after each polysomnography measurement in order to closely and prospectively monitor and describe potential changes in their sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Poul Jennum, Professor, Study Director — Danish center for sleep medicine, department of clinical neurophysiology, Glostrup Hospital, Copenhagen University, Denmark
Locations (1):
- Glostrup Hospital, Copenhagen University, Glostrup Municipality, Copenhagen, Denmark

REFERENCES:
- [Derived] Loppenthin K, Esbensen BA, Jennum P, Ostergaard M, Christensen JF, Thomsen T, Bech JS, Midtgaard J. Effect of intermittent aerobic exercise on sleep quality and sleep disturbances in patients with rheumatoid arthritis - design of a randomized controlled trial. BMC Musculoskelet Disord. 2014 Feb 21;15:49. doi: 10.1186/1471-2474-15-49. PMID 24559487